CLINICAL TRIAL: NCT06482970
Title: Brain Function, Clinical and Psychosocial Outcomes After Neuromuscular Exercise Plus Pain Neuroscience Education Intervention in Patients With Chronic Pain Due to Knee Osteoarthritis. A Randomized Controlled Trial Protocol
Brief Title: Effectiveness of Exercise Plus Pain Neuroscience Education on Brain Function in Knee Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Santo Tomas, Chile (Other)
Responsible Party: Principal Investigator, Joaquín Ignacio Salazar Méndez, principal investigator, Universidad Santo Tomas, Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-02
Record Dates: First submitted 2024-06-20; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Knee Osteoarthritis
Keywords: Neuromuscular exercise; Pain neuroscience education; Knee osteoarthritis; Chronic pain; Physical therapy
MeSH Terms: conditions — Osteoarthritis, Knee; Chronic Pain | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neuromuscular exercise plus Pain neuroscience education (Experimental): Neuromuscular exercise will be carried out for eight weeks, with three weekly sessions, in groups (up to five participants per group).
  Each session will consist of three parts: warm-up, exercise circuit and cool down. Each part will be regulated for the abilities of the participants
  Pain neuroscience education will be carried in group using visual support for Powerpoint presentations. The PNE will include five dimensions with a focus on reducing fear-avoidance beliefs and catastrophic thoughts to promote self-efficacy. Five PNE sessions will be carried out, one for each dimension, with a duration of 30-45 minutes each taught during the first five sessions of the intervention. In addition, a brochure will be delivered with the main points of each of the domains and an informative video will be made to which participants will have access (five 15-minute videos, one per domain).
  Interventions: Other: Neuromuscular exercise plus pain neuroscience education
- Neuromuscular exercise (Experimental): Neuromuscular exercise will be carried out for eight weeks, with three weekly sessions, in groups (up to five participants per group).
  Each session will consist of three parts: warm-up, exercise circuit and cool down. Each part will be regulated for the abilities of the participants
  Interventions: Other: Neuromuscular exercise
- Usual care (No Intervention): Participants will be urged to continue with their life activities without changes. All participants will continue to receive routine care offered by their doctor and other health care providers. No trial interventions were provided. The possible treatments that may be provided to the participants in this group (if the primary medical team deems it appropriate) will not be influenced. However, if the participants receive any treatment from their medical staff, it will be recorded as an extra history and the participant will not be considered in the analyses. All participants in this group will be eligible to receive the experimental therapies of their choice once the study is completed.

INTERVENTIONS:
Other: Neuromuscular exercise plus pain neuroscience education — The exercises follow neuromuscular principles, which aim to improve sensorimotor control and achieve compensatory functional stability (also called dynamic stability).
  Pain neuroscience education will take an active, person-centered approach through their own fear-avoidance beliefs.
  Arms: Neuromuscular exercise plus Pain neuroscience education
Other: Neuromuscular exercise — The exercises follow neuromuscular principles, which aim to improve sensorimotor control and achieve compensatory functional stability (also called dynamic stability).
  Arms: Neuromuscular exercise

SUMMARY:
A three-arm randomized controlled trial will be conducted. Fifty-nine participants with KOA will be recruited in a 1:1:1 ratio. Assessor, and statistician will be blinded to group allocation. One experimental group (n=19) will receive NME plus PNE, the other experimental group (n=19) will receive isolated NME and the control group (n=19) will continue with usual care. The PNE will be adapted to the context of the participants. Outcome measures will be brain activity, pressure pain threshold, pain intensity, disability, fear-avoidance beliefs, self-efficacy, and pain catastrophizing. Outcome measures will be evaluated pre-intervention, immediately post-intervention, and four-month post-intervention.

The investigators hypothesize that there will be significant differences in favor of the NME plus PNE intervention group.

ELIGIBILITY:
Inclusion Criteria:

* women and men at least 45 years old radiologically diagnosed with unilateral or bilateral KOA (Kellgren-Lawrence 1-3 grading scale)
* pain duration greater than three months

Exclusion Criteria:

* Patients who have received physical therapy or other conservative therapy in the previous three months and those who have a history of major knee trauma and surgery in the last six months
* cardiac pathology
* structural use of psychoactive medications, such as antipsychotics, antidepressants, antiepileptics, and anxiolytics, during the past year
* neurological diseases
* other musculoskeletal clinical conditions that generate pain

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Brain function (peak frequency) | baseline, post-intervention (2 months after admission), follow-up four months after the intervention.
  An analysis of the peak frequencies (the highest power frequency determined in the average of the windows as the local maximum (greater than its two neighboring windows) of the amplitude in a frequency range of 6-14 Hz will be applied.
Brain function (power spectrum) | baseline, post-intervention (2 months after admission), follow-up four months after the intervention.
  A global analysis of the power spectrum will be carried out, considered as the average of all the electrodes, which represents the synchronization between the neurons to generate the discharges. A topographic power analysis will also be performed for the Delta (0.1 - 4 Hz), theta (4 - 8 Hz), alpha (8 - 13 Hz) and beta (13 - 30 Hz) frequency bands.

SECONDARY OUTCOMES:
Pain pressure-threshold | baseline, post-intervention (2 months after admission), follow-up four months after the intervention.
  A digital algometer (WAGNER FDX10) will be used to measure pressure pain sensitivity. The average of three measurements will be used. Patients will be evaluated lying supine in a comfortable position according to the area to be evaluated. It will be performed at two test sites on the affected knee(s) (3 cm medial and lateral to the midpoint of the medial and lateral edge of the patella, respectively) and will also be applied to a distant site on the ipsilateral carpal extensor radialis longus (5 cm distal to the lateral epicondyle).
Pain intensity | baseline, post-intervention (2 months after admission), follow-up four months after the intervention.
  The pain intensity will be measured with the Visual Analogue Scale (VAS), which consists of a 10 cm straight line with two labels, at one end "no pain" and at the other "the worst possible pain" where the patient will draw a vertical mark indicating your pain level. The pain intensity at rest and during activity in the last 7 days will be considered.
Disability | baseline, post-intervention (2 months after admission), follow-up four months after the intervention.
  Disability will be assessed with the Western Ontario and McMaster Universities Osteoarthritis (WOMAC) questionnaire. It consists of 24 questions divided into 3 domains: pain, stiffness and physical function with 5, 2 and 17 questions, respectively. Each question is scored on a Likert scale of 0-4, corresponding to the intensity levels of none, slight, moderate, severe and extreme pain. A higher WOMAC score indicates worse health status.
Fear-avoidance beliefs | baseline, post-intervention (2 months after admission), follow-up four months after the intervention.
  Fear-avoidance beliefswill be evaluated with the Fear Avoidance Beliefs Questionnaire (FABQ). This questionnaire consists of 2 subscales with 16 items in total 70. It is rated on a 7-point Likert scale (0=strongly disagree to 6=strongly agree).
Self-efficacy | baseline, post-intervention (2 months after admission), follow-up four months after the intervention.
  Self-efficacy will be evaluated with the Pain Self-Efficacy Questionnaire (PSEQ) will be used. It consists of 10 items rated on a 7-point Likert scale from 0 ("not at all confident") to 6 ("very confident")
Pain Catastrophizing | baseline, post-intervention (2 months after admission), follow-up four months after the intervention.
  Pain catastrophizing will be assessed using the Pain Catastrophizing Scale (PCS) questionnaire. It consists of 3 subscales (rumination, magnification and helplessness) with 13 questions in total, which are scored on a Likert scale from 0 (mild symptoms) to 4 (worst symptoms) points. The higher the score, the more pain catastrophizing the patient presents.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquín I Salazar, MSc, Principal Investigator — Universidad Santo Tomás

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: from 6 months after publication. They will be available for one year
Access Criteria: will be provided to any researcher who requires it via email